CLINICAL TRIAL: NCT01412528
Title: Phase II Study to Standardize Allergen Extracts: Determination of Biological Activity in HEP Units
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: University of Zurich (Other)
Responsible Party: Kuendig Thomas Dr., University hospital Zurich, Dermatology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZU-EASY-001
Record Dates: First submitted 2010-04-28; First posted 2011-08-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-01

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

ARMS (1):
- Eight different allergens will be standardized in this study (Other)
  Interventions: Other: Allergen extracts

INTERVENTIONS:
Other: Allergen extracts

SUMMARY:
Today a variety of diagnostic tools to detect allergenic agents are available such as skin tests, provocation tests and blood tests. Due to its high sensitivity and low costs the skin prick test is the most commonly used test to identify allergies in patients. By using this kind of skin test, up to 25 different agents can be tested in parallel, rendering the skin prick test a cheap, easy-to-handle and rapid diagnostic tool. However, as research proceeds, new tools appear with the intention to make future applications even more convenient -for both, the patient and the physician. For that purpose the development of the so called "Easyprick" Allergen Test System is under way, consisting of a foil that carries ready-to-use, allergen-soaked sponges which can easily be applied to the skin after pricking.

Allergen extracts are complex mixtures of proteins and contain varying amounts of allergenic and non-allergenic components. In order to control variability and to achieve consistency and reproducibility for optimal safety and sensitivity/specificity, it is essential to standardize the amount of allergen used in prick tests. The present study aims to standardize eight allergen extracts by using this method. Standardized extracts will then be applied in the Easyprick Allergen Test System which will be evaluated and compared to the conventional prick test in a second study.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* 18-65 years old,
* a positive clinical history for inhalant allergy to at least one of the allergens to be tested,
* at least one positive prick test (mean wheal diameter = 3mm) when tested with already standardized extracts of the allergens under investigation.
* a mean wheal size of = 7mm2 obtained in a prick test with histamine dihydrochloride (10mg/ml).
* Written informed consent

Exclusion criteria: -currently suffering from allergy symptoms,

* history of systemic reactions to allergens,
* severe diseases influencing the results of the present study by discretion of the investigator,
* immunotherapy with an allergen preparation known to interfere with the allergens under investigation during the past two years,
* skin lesions in the skin test areas
* pregnancy or nursing,
* treatment with prohibited concomitant medications (antihistamines, corticosteroids, anti-depressants, neuroleptics or specific immunotherapy)
* alcohol or drug abuse,
* impaired in understanding nature, meaning and the scope of the study or are incapable of giving written informed consent,
* Participation in another clinical trial within the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Wheal size
  15 minutes after skin prick test with a serial dilution of an allergen extracts, sizes of provoked wheals will be measured according to allergen standardization procedure.

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Clinical Trials Center, Zurich, Switzerland